CLINICAL TRIAL: NCT06166472
Title: A Phase I Study to Evaluate the Safety, Tolerance, Pharmacokinetics, and Preliminary Antineoplastic Activity of The Anti-CLDN18.2 and CD47 Bispecific Antibody AK132 in Advanced Malignant Solid Tumor
Brief Title: A Study to Evaluate the Safety, Tolerance, Pharmacokinetics, and Preliminary Antineoplastic Activity of AK132 in Advanced Malignant Solid Tumor
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK132-101
Record Dates: First submitted 2023-11-23; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Advanced Malignant Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK132 (Experimental): Each subject will receive a single dose of AK132 every 2-week cycle (Q2W).
  Interventions: Drug: AK132

INTERVENTIONS:
Drug: AK132 — IV infusion, specified dose on specified days.

SUMMARY:
This is A Phase I Study to Evaluate the Safety, Tolerance, Pharmacokinetics, and Preliminary Antineoplastic Activity of The anti-CLDN18.2 and CD47 Bispecific Antibody AK132 in Advanced Malignant Solid Tumor

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the study with full informed consent and signed written informed consent form.
2. Males or females aged ≥ 18 to ≤ 75 years at the time of signing informed consent.
3. Histologically and/or cytologically confirmed locally advanced unresectable or metastatic malignant solid tumors.
4. The interval between the end of the last systemic anti-tumor treatment and the first dose should be at least 3 weeks.
5. Subjects in the dose expansion phase are required to provide tumor tissue samples.
6. At least one measurable tumor lesion per RECIST v1.1.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Life expectancy ≥ 3 months.
9. Adequate organ function as assessed in the laboratory tests.
10. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose and agree to take effective contraception measures during the study drug administration and within 120 days after the last dose. Male patients with female partners of childbearing potential must agree to take effective contraception measures during the study drug administration and within 120 days after the last dose.

Exclusion Criteria:

1. There is active or untreated brain metastases,Meningeal metastases, spinal cord compression, or leptomeningeal disease.
2. Presence of clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring frequent drainage (≥ 1/month).
3. Patients who, in the opinion of the investigator, have symptoms or signs suggestive of clinically unacceptable deterioration of the primary disease at the time of screening.
4. gastrointestinal perforation or gastrointestinal fistula within 6 months before the first dose.
5. clinically significant bleeding symptoms or a clear tendency to bleed within 4 weeks before the first dose.
6. Active malignant tumors within the past 3 years, except for tumors in this study and scured local tumors.
7. History of hemolytic anemia due to any cause within 3 months before the first dose of study drug.
8. Have a history of defects in red blood cell or hemoglobin production or metabolism.
9. Major surgery other than the diagnosis of solid tumors within 28 days prior to the first dose or major surgery is expected during the study.
10. Clinically significant cardiovascular or cerebrovascular disease.
11. Presence of ≥ Grade 2 peripheral neuropathy as defined by NCI CTCAE v5.0.
12. Presence of active diverticulitis.
13. Patients with serious neurological or psychiatric disorders.
14. Pregnant or lactating women.
15. Patients who received palliative local therapy for any tumor lesions within 2 weeks prior to the first dose;and Chinese herbal medicine or traditional Chinese medicinal products with anti-tumor indications within 2 weeks prior to the first dose.
16. Serious adverse reactions in subjects who have previously received anti-PD-1/PD-L1/CTLA-4 or any other immunotherapy or immuno-oncology (IO) drug.
17. Patients who require systemic treatment with glucocorticoids (> 10 mg/day prednisone or equivalent) or other immunosuppressive drugs within14 days prior to the first dose.
18. Unresolved toxicities during prior anti-tumor therapy with the exception of alopecia/pigmentation.
19. Subjects with a known history of severe hypersensitivity to other monoclonal antibodies. A known history of allergy or hypersensitivity to AK132 or any of its components.
20. Previous use of any antineoplastic drug targeting the CD47-SIRPα pathway or Claudin18.2.
21. Active autoimmune disease requiring systemic treatment within 2 years prior to the start of study treatment, or autoimmune diseases that may relapse or require scheduled treatment as judged by the Investigator.
22. Known active pulmonary tuberculosis.
23. Patients with active hepatitis B or active hepatitis C.
24. Known medical history of immunodeficiency or positive HIV test.
25. Known presence of interstitial lung disease or noninfectious pneumonitis that is currently symptomatic or requires prior systemic glucocorticoid therapy that, in the judgment of the Investigator, may affect the assessment or management of toxicity related to study treatment.
26. Patients with active infection, including those requiring intravenous antibiotics or antifungal therapy for 2 weeks prior to first dose, and unexplained fever during screening (CTCAE≥1, except those determined by the investigator to be neoplasmic).
27. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
28. Live vaccines were administered within 28 days prior to the first dose or were planned to be administered during the study period.
29. Concurrent participation in another clinical study, unless it is an observational, non-interventional clinical study or the follow-up period of an interventional study.
30. Any condition that, in the opinion of the Investigator, may result in a risk when receiving the study drug, or would interfere with the evaluation of the study drug or the safety of patients, or the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-12-12 (Estimated); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicity （DLT）、adverse event（AE）、serious adverse event（SAE） | Up to 2 years
  incidence and severity of DLT, adverse events (AE), serious adverse events (SAE)
Maximum tolerated dose (MTD),RP2D | Up to 2 years
  Maximum tolerated dose (MTD), Recommended dose for phase II trial

SECONDARY OUTCOMES:
Pharmacokinetic | Up to 2 years
  The PK parameters include serum concentrations of AK132 at different timepoints after AK132 administration.
Immunogenicity assessmen | Up to 2 years
  The immunogenicity of AK132 will be assessed by summarizing the number and percentage of subjects who develop detectable antidrug antibodies (ADAs).
Objective response rate (ORR) | Up to 2 years
  ORR is the proportion of subjects with CR or PR based on RECIST v1.1
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST Version 1.1) or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (based on RECIST Version 1.1).
Time to response (TTR) | Up to 2 years
  Time to response (TTR) is defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieved CR or PR (based on RECIST Version 1.1).
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST Version 1.1).
Overall survival (OS) | Up to 2 years
  OS defined as the time from the first dose to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, M.D., Principal Investigator — Name:Sun Yat-Sen University Cancer Center, Guangzhou, China
Locations (7):
- China (7):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, China, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Huazhong University of Science and Technology Tongji Medical College Affiliated Union Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Provincial Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No